CLINICAL TRIAL: NCT04965194
Title: Ultrasound-guided Erector Spinae Block Versus Quadratus Lumborum Block for Postoperative Analgesia in Laparotomies: Randomized Controlled Study
Brief Title: Ultrasound-guided Erector Spinae Block Versus Quadratus Lumborum Block for Laparotomies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Shadwa Rabea Mohamed, lecturer, Minia University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 50:6/2021
Record Dates: First submitted 2021-07-03; First posted 2021-07-16 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-11

CONDITIONS: Analgesia
Keywords: ESPB; QLPB; analgesia; postoperative pain
MeSH Terms: conditions — Agnosia; Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Erector spinae plane block (ESPB) (Experimental): 20 ml of 0.25% bupivacaine will be administered to perform ESP block on each side
  Interventions: Procedure: erector spinae plane block
- Quadratus lumborum plane block (QLPB) (Experimental): The injectate (20ml of bupivacaine 0.25%) should ideally spread from the injection site inside the fascial plane between the QL and psoas major muscles to the thoracic paravertebral space with a goal to accomplish segmental somatic and visceral analgesia from T4 to L1.
  Interventions: Procedure: Quadratus lumborum plane block
- Control group (Placebo Comparator): patients received no regional block
  Interventions: Other: placebo

INTERVENTIONS:
Procedure: erector spinae plane block — Superficial probe will be placed 2-3 cm lateral to the spine using a sagittal approach at the level of T8. After identification of erector spinae muscle and transverse processes, the needle will be inserted deeply into the erector spinae muscle. Correct position of the needle tip is confirmed with administration of 0.5-1 ml of local anesthetic (LA), and 20 ml of 0.25% bupivacaine will be administered to perform ESP block. LA spread to both cranial and caudal directions will be seen.
  Arms: Erector spinae plane block (ESPB)
Procedure: Quadratus lumborum plane block — A curved array transducer for the transmuscular QL (TQL) nerve block is placed in the axial plane on the patient's flank just cranial to the iliac crest. The "shamrock sign" is visualized: The transverse process of vertebra L4 is the stem, whereas the erector spinae posteriorly, QL laterally, and psoas major anteriorly represents the three leaves of the trefoil. The target for injection is the fascial plane between the QL and psoas major muscles. The needle is inserted using an in-plane technique from the posterior end of the transducer through the QL muscle. The injectate (20ml of bupivacaine 0.25%) should ideally spread from the injection site inside the fascial plane between the QL and psoas major muscles to the thoracic paravertebral space with a goal to accomplish segmental somatic and visceral analgesia from T4 to L1.
  Arms: Quadratus lumborum plane block (QLPB)
Other: placebo — patients received no regional block
  Arms: Control group

SUMMARY:
The study aimed to compare the effect of ESP block and QL block in preventing postoperative pain and decreasing analgesic consumption in patients scheduled for laparotomies.

This prospective randomized controlled study will be done after obtaining ethics committee's permission and written informed consent of the patients 60 adult patients aged 18-60 years scheduled for open laparotomies under general anesthesia will be included in this study.

According to the used technique, the patients will be randomly allocated into 3 parallel equal groups (20 patients in each one).

Group I (ES group): the patients will receive bilateral ESP block. Group II (QL group): the patients will receive bilateral QL block. Group III (control group): the patients will not receive any regional block.

DETAILED DESCRIPTION:
Postoperative pain management is one of the most important issues influencing the outcome of surgery. Postoperative pain, especially when poorly controlled, results in harmful acute effects such as adverse physiological responses and chronic effects like delayed long term recovery and chronic pain.the investigators aimed to compare the effect of ESP block and QL block in preventing postoperative pain and decreasing analgesic consumption in patients scheduled for laparotomies.

Primary outcome:

Total analgesic consumption in the first 24hrs postoperative.

Secondary outcomes:

1. Time of first analgesic request.
2. Visual analogue pain score in the first 24hrs postoperative
3. Incidence of any side effects. All patients will be premedicated using midazolam 0.03 mg /kg iv upon arrival to the operating room then standard monitoring which included SPO2, ECG, non-invasive blood pressure monitoring will be applied. All patients will receive the same anesthetic technique. Following anesthesia induction using 1-2 mcg/kg fentanyl, 2- 3 mg/kg propofol, and 0.5 mg/kg atracurium, the patients will be intubated and maintenance of anesthesia will be done by Isoflurane (MAC 1.2) and intermittent doses of atracurium to maintain adequate muscle relaxation. All hemodynamics will be measured before and after induction of general anesthesia and then every 5 min till end of surgery.

In ES group: superficial probe will be placed 2-3 cm lateral to the spine using a sagittal approach at the level of T7. After identification of erector spinae muscle and transverse processes, the needle will be inserted deeply into the erector spinae muscle. Correct position of the needle tip is confirmed with administration of 0.5-1 ml of local anesthetic (LA), and 20 ml of 0.25% bupivacaine will be administered to perform ESP block. LA spread to both cranial and caudal directions will be seen.

In QL group: A curved array transducer for the transmuscular QL (TQL) nerve block is placed in the axial plane on the patient's flank just cranial to the iliac crest. The "shamrock sign" is visualized: The transverse process of vertebra L4 is the stem, whereas the erector spinae posteriorly, QL laterally, and psoas major anteriorly represents the three leaves of the trefoil. The target for injection is the fascial plane between the QL and psoas major muscles. The needle is inserted using an in-plane technique from the posterior end of the transducer through the QL muscle. The injectate (20ml of bupivacaine 0.25%) should ideally spread from the injection site inside the fascial plane between the QL and psoas major muscles to the thoracic paravertebral space with a goal to accomplish segmental somatic and visceral analgesia from T4 to L1.

Before the end of the surgery all patients will receive 1g of paracetamol IV, at the end of the surgery reversal of neuromuscular blockade will be done by neostigmine and atropine and then the patients will be transferred to recovery room. 30 mg of ketorolac will be given to all patients every 8 hrs.

Parameters will be assessed:

Intraoperative:

Hemodynamics after induction of anesthesia, after block and then every 15min till the end of surgery.

Postoperative:

1. Hemodynamics immediately after recovery and then 1, 2, 4, 8, 12, 16, 20and 24 hrs postoperative.
2. VAS in the same previous intervals.
3. Time of first analgesic request.
4. Total analgesic requirement in the first 24 hrs. postoperative.
5. Incidence of side effects.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-60 years.
* ASA I-II.
* Both sexes.
* Open laparotomies.

Exclusion Criteria:

1. Patient refusal
2. Allergy to local anesthetics
3. BMI >40 kg/m2
4. Bleeding diathesis or history of anticoagulant use.
5. Psychiatric diseases.
6. Infection of the skin at the site of needle punctures area.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2021-07-15 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
Total analgesic consumption | 24 hours
  total fentanyl consumption as rescue analgesia

SECONDARY OUTCOMES:
Time of first analgesic request. | 24 hours
  first dose of rescue analgesia
dynamic Visual analogue pain score | 24 hours
  degree of pain description on movement from (0-10 )which 0-3 is the no pain, 4-5 mild pain, 6-8 moderate pain and 9-10 severe pain
resting Visual analogue pain score | 24 hours
  degree of pain description on rest from (0-10 )which 0-3 is the no pain, 4-5 mild pain, 6-8 moderate pain and 9-10 severe pain

CONTACTS AND LOCATIONS:
Overall Officials: Shadwa R Mohamed, MD, Study Chair — Mina university hospital; Ahmed H Mohamed, Study Director — Minia Universiry hospital
Locations (1):
- Minia University Hospital, Minya, Minya Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No